CLINICAL TRIAL: NCT06649409
Title: An Open-label, Randomized, 3-arm, Parallel-group, Positive- and Negative-arm Controlled Study to Evaluate the Mineralocorticoid Receptor Antagonism Effect of Vamorolone in Healthy Subjects
Brief Title: Evaluation of Vamorolone Mineralocorticoid Receptor Antagonism in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Santhera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SNT-I-VAM-026; 2024-512101-60-00 (EU CTIS Number); N-A-PH1-23-067 (Other: Nuvisan)
Record Dates: First submitted 2024-09-05; First posted 2024-10-18 (Actual); Results first posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Pharmacodynamic
Keywords: Mineralocorticoid Receptor Antagonism
MeSH Terms: interventions — VBP15 compound; Drugs, Investigational; Eplerenone; Fludrocortisone

STUDY DESIGN:
Intervention Model Description: This study will be conducted in a single-center, randomized, open-label, 3-arm, parallel-group, positive- and negative-controlled design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Study arm 1 vamorolone (Experimental): Vamorolone 20 mg/kg single dose on Day 2 and Fludrocortisone challenge on Days 1 to 3
  Interventions: Drug: Vamorolone; Drug: Fludrocortisone
- Study arm 2 (positive control arm): eplerenone (Active Comparator): Eplerenone 200 mg single dose on Day 2 and Fludrocortisone challenge on Days 1 to 3
  Interventions: Drug: Eplerenone; Drug: Fludrocortisone
- Study arm 3 (negative control arm): no "active" treatment (Other): Fludrocortisone challenge on Days 1 to 3
  Interventions: Drug: Fludrocortisone

INTERVENTIONS:
Drug: Vamorolone — vamorolone 20 mg/kg single dose on Day 2
  Other Names: experimental drug
  Arms: Study arm 1 vamorolone
Drug: Eplerenone — Eplerenone 200 mg single dose on Day 2
  Other Names: positive control
  Arms: Study arm 2 (positive control arm): eplerenone
Drug: Fludrocortisone — Fludrocortisone challenge on Days 1 to 3 (for all subjects):
  Day 1:
  -Fludrocortisone 1 mg at 9 h predose vamorolone /eplerenone administration/corresponding timepoint for negative control arm
  Day 2:
  * Fludrocortisone 0.5 mg at the same time of vamorolone/eplerenone administration in the morning (0 h) /corresponding timepoint for negative control arm.
  * Fludrocortisone 0.1 mg at 2 h, 4 h, 6 h, 8 h, 10 h, 12 h, and 14 h vamorolone/eplerenone postdose administration/corresponding timepoint for negative control arm.
  * Fludrocortisone 0.5 mg at 16 h vamorolone/eplerenone postdose administration/corresponding timepoint for negative control arm.
  Day 3:
  -Fludrocortisone 0.1 mg at 24 h vamorolone/eplerenone postdose administration on Day 2/corresponding timepoint for negative control arm.
  Other Names: auxiliary medicinal product - mineralocorticoid agonist

SUMMARY:
To evaluate if the trial drug vamorolone is able to block a specific receptor in the body called mineralocorticoid receptor. This receptor helps to regulate salt and water balance.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the antagonistic effect of vamorolone on the mineralocorticoid receptor following mineralocorticoid challenge by fludrocortisone, compared to eplerenone as a positive control, and to a negative control with no study treatment. Furthermore, the safety and tolerability of vamorolone combined with fludrocortisone challenge will be assessed, and the Pharmacokinetic (PK) of a single dose of vamorolone and a single dose of eplerenone, combined with fludrocortisone challenge, will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 to 55 years inclusive, at the time of signing the informed consent.
2. Male is overtly healthy as determined by medical evaluation including medical history, physical examination, vital signs, laboratory tests and ECG.
3. Body weight ≥ 50 kg and a BMI ≥ 18 kg/m2 and ≤ 29.9 kg/m2 at screening
4. Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

   If the subject is a sexually active man and not surgically sterilized, he must be willing to:
   * Abstain from sexual intercourse or
   * Use a condom plus another form of contraception (e.g., spermicide, Intrauterine device (IUD), birth control pills taken by female partner, diaphragm with spermicide) if engaging in sexual intercourse with a woman who could become pregnant.
   * Use a condom during sexual intercourse with pregnant or lactating women.
   * Must not father a child and must refrain from donating sperm from administration of the first dose and up to 3 months after the last dose of study treatment.
5. Subject is a non-smoker for at least 3 months prior to exposure to the study treatments.

   Subjects must also have abstained from use of other nicotine containing products (e.g., nicotine patch, chewing gum or e-cigarettes) for at least 3 months before exposure to the study treatment.
6. Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the Informed consent form (ICF) and in this protocol prior to any clinical study specific procedure.
7. Supine systolic blood pressure of ≥ 90 mmHg and ≤ 140 mmHg, diastolic blood pressure of ≥ 50 mmHg and ≤ 90 mmHg, pulse rate of ≥ 45 bpm and ≤ 90 bpm, and tympanic body temperature of ≥ 35.0 and ≤ 37.5°C at screening.
8. Subjects must be able to communicate well with the Investigator and comply with the protocol requirements, instructions, and protocol related restrictions (e.g., dietary, fluid and lifestyle restrictions from screening to study completion)
9. Subjects must be able to swallow the study treatments as per protocol

Exclusion Criteria:

1. A past medical history of clinically significant abnormalities or a history/family history of long QT interval syndrome.
2. An abnormal ECG, defined as:

   * Pulse rate (PR) > 215 msec and < 120 msec, QRS (Part of electrocardiographic wave representing ventricular depolarization) complex > 120 msec; QTcF > 440 msec by automated reading
   * Any clinically significant cardiac conduction abnormalities
   * Any atrial or ventricular arrhythmias
3. A past medical history of myocardial infarction, angina pectoris, atherosclerosis, or other clinically significant heart disease (e.g.congestive heart failure, uncontrolled hypertension, history of labile hypertension)
4. A past medical history of peptic ulcers, diverticulitis, and non-specific ulcerative colitis.
5. History of complaints of frequent dizziness and /or vomiting spells or lightheadedness.
6. Any history or evidence of any clinically relevant, gastrointestinal, respiratory, hepatic, renal, endocrinologic, hematologic, immunologic, metabolic, genitourinary, pulmonary, neurologic, dermatologic, musculoskeletal, and/or other major disease or malignancy as determined by medical evaluation (including physical examination) capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study treatments; or interfering with the interpretation of data.
7. Known Gilbert's syndrome.
8. Any clinically relevant history of allergic conditions requiring hospitalization or prolonged systemic treatment (including drug allergies, allergic asthma, eczema, allergies requiring therapy with corticosteroids or anaphylactic reactions); but excluding untreated, asymptomatic, seasonal allergies at time of dosing or allergic contact sensitizations (e.g., nickel allergy).
9. Known or suspected hypersensitivity or contraindications to the study treatments or any components of the formulation used, e.g., vamorolone, eplerenone and fludrocortisone.
10. Relevant current acute or chronic/recurrent viral, bacterial, fungal or parasitic infections (e.g., pulmonary/upper respiratory, gastrointestinal, urinary, skin, or ear, nose and throat (ENT) infections) at screening or within 28 days prior to administration of the study treatments.
11. Use of any concomitant medication or any drugs / medicines (including dietary supplements, natural and herbal remedies, and hormone replacement therapy) within 2 weeks or 5 times the half-life of the respective drug, whichever is longer, prior to the first administration of the study treatments.

    Occasional use of paracetamol up to 2 g/day (medicinal product in its original packaging, approved and marketed in Germany) is permitted.

    Oral, injectable, and implantable contraceptives as outlined in protocol section 5.1 are permitted.
12. Previous exposure to vamorolone.
13. Any use of corticoids within 6 months prior to the first administration of the study treatments.
14. Administration of live, attenuated, replication-competent vaccines within 6 weeks prior to the first administration of study treatment until 2 weeks after the follow-up visit. Administration of inactivated vaccines or vector-based or messenger ribonucleic acid (mRNA ) COVID-19 vaccines within 2 weeks prior to the first administration of the study treatments until 2 weeks after the follow-up visit.
15. Treatment with biologic agents (such as monoclonal antibodies including marketed drugs) within 3 months or 5 half-lives (whichever is longer) prior to the first administration of the study treatments.
16. Use of any investigational drug or participation in any clinical study within 30 days or 5 half-lives (whichever is longer) prior to the expected date of first administration of study treatments or planning to take other investigational drugs during the study.
17. Positive results for HBsAg, anti-HCV (Hepatitis C virus), anti-HIV 1 and 2, and HIV 1-p24 antigen at screening.
18. Positive screen for alcohol, drugs of abuse and cotinine at screening.
19. Elevations in Alanine aminotransferase (ALT) ≥ 1.1 x ULN (Upper limit of normal) , AST (Aspartate aminotransferase) ≥ 1.1 x ULN, serum bilirubin ≥ 1.0 x ULN, creatinine ≥1.0 x ULN and HbA1c > ULN at screening. A case-by-case decision for any abnormality must be discussed with the Sponsor before inclusion.
20. Sodium, potassium, magnesium, chloride blood concentration below the lower limit of normal at screening.
21. Thyroid-stimulating hormone (TSH) and coagulation outside of normal ranges.
22. eGFR (Estimated glomerular filtration rate) based on the Chronic kidney disease epidemiology collaboration (CKD-EPI) of < 90 mL/min at screening.
23. Subjects who are unwilling to adhere to contraceptive requirements.
24. Higher than low-risk alcohol consumption i.e., consumption of an average weekly alcohol intake of > 21 units/week for men. 1 unit (12 g) corresponds to 0.3 L of beer/day or 0.12 L of wine/day or 1 glass (at 2 cL) of spirits/day.
25. Excessive consumption of caffeine- or xanthine-containing food or beverages (> 5 cups of coffee a day or equivalent) or inability to stop consuming from 48 hours prior to first planned administration of study treatments.
26. Consumption of alcohol from 48 hours prior to admission
27. Consumption of high-dose resveratrol-containing products or products with enzyme-inducing or enzyme-inhibiting properties 14 days prior to first administration of study treatments.
28. Regular consumption of poppy seed containing food prior to first administration of study treatments.
29. No sweets/teas containing liquorice are allowed within 2 weeks prior to first administration of study treatments up to the follow-up examination.
30. Any use of drugs-of-abuse or alcohol abuse within 1 month prior to dosing.
31. Subject with vegetarian, vegan, or restricted diet (e.g., gluten-free) or not willing or able to eat the complete standard meals.
32. Donation or loss of more than 400 mL of blood or received a transfusion of any blood or blood products within 30 days, or donated plasma within 30 days prior to first administration of study treatments.
33. Strenuous physical activity within 72 h to admission.
34. Employee of the Sponsor, the Nuvisan Group, or other Contract Research Organization involved in the clinical study.
35. Legal incapacity or limited legal capacity, or incarceration and vulnerable subjects.
36. Inability to understand or communicate reliably with the Investigator or considered by the Investigator to be unable to or unlikely to co-operate with the protocol requirements, instructions, and study-related restrictions
37. History of non-compliance to medical regimens and subjects who are considered potentially unreliable (e.g., refuse to comply with study regulations).
38. Any other conditions or factors which in the opinion of the Investigator may interfere with study conduct.
39. Changes in medical conditions compared to screening, as judged by the Investigator.
40. Body weight < 50 kg.
41. Changes in prior/concomitant therapy compared to screening, as judged by the Investigator.
42. Positive for an acute common cold/respiratory or other infection upon admission.
43. Positive screen for alcohol, drugs of abuse and cotinine test upon admission.
44. Changes in other exclusion criteria compared to screening, as judged by the Investigator.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-06-05 (Actual); Primary Completion 2024-06-29 (Actual); Study Completion 2024-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Haffner, MD, Principal Investigator — Nuvisan GmbH
Locations (1):
- Nuvisan GmbH, Neu-Ulm, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] de Vera A, Clemens PR, Dang UJ, Dutreix C, Gresko E, Guglieri M, Hagerty L, Hasham S, Damsker J, Hathout Y, Linden A, Berglund A, Tobin R, Wahbi K, Hoffman EP. Mineralocorticoid receptor antagonism of vamorolone: Evidence from LIONHEART and VISION-DMD clinical trials. Steroids. 2025 Nov;223:109689. doi: 10.1016/j.steroids.2025.109689. Epub 2025 Sep 14. PMID 40957504

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Arm 1 (Test Arm)Vamorolone: single oral dose of vamorolone 20 mg/kg on day 2
  + Fludrocortisone Challenge Day 1: 1 mg single dose at 9 h predose vamorolone dosing. Day 2: 0.1 mg and 0.5 mg multiple doses. For detailed timepoints, see protocol Section 4.1. Day 3: 0.1 mg single dose at 24 h postdose vamorolone dosing.
  Vamorolone: vamorolone 20 mg/kg single dose on Day 2
  Fludrocortisone: Fludrocortisone challenge on Days 1 to 3 (for all subjects):
  Day 1:
  -Fludrocortisone 1 mg at 9 h predose vamorolone /eplerenone administration/corresponding timepoint for negative control arm
  Day 2:
  * Fludrocortisone 0.5 mg at the same time of vamorolone/eplerenone administration in the morning (0 h) /corresponding timepoint for negative control arm.
  * Fludrocortisone 0.1 mg at 2 h, 4 h, 6 h, 8 h, 10 h, 12 h, and 14 h vamorolone/eplerenone postdose administration/corresponding timepoint for negative control arm.
  * Fludrocortisone 0.5 mg at 16 h vamorolone/eplerenone postdose administration/corresponding timepoint for negative control arm.
  Day 3:
  -Fludrocortisone 0.1 mg at 24 h vamorolone/eplerenone postdose administration on Day 2/corresponding timepoint for negative control arm.
- Study Arm 2 (Positive Control Arm): Eplerenone: single oral dose of eplerenone 200 mg on day 2
  + Fludrocortisone challenge Day 1: 1 mg single dose at 9 h predose eplerenone dosing. Day 2: 0.1 mg and 0.5 mg multiple doses. For detailed timepoints, see protocol Section 4.1. Day 3: 0.1 mg single dose at 24 h postdose eplerenone dosing.
  Eplerenone: Eplerenone 200 mg single dose on Day 2
  Fludrocortisone: Fludrocortisone challenge on Days 1 to 3 (for all subjects):
  Day 1:
  -Fludrocortisone 1 mg at 9 h predose vamorolone /eplerenone administration/corresponding timepoint for negative control arm
  Day 2:
  * Fludrocortisone 0.5 mg at the same time of vamorolone/eplerenone administration in the morning (0 h) /corresponding timepoint for negative control arm.
  * Fludrocortisone 0.1 mg at 2 h, 4 h, 6 h, 8 h, 10 h, 12 h, and 14 h vamorolone/eplerenone postdose administration/corresponding timepoint for negative control arm.
  * Fludrocortisone 0.5 mg at 16 h vamorolone/eplerenone postdose administration/corresponding timepoint for negative control arm.
  Day 3:
  -Fludrocortisone 0.1 mg at 24 h vamorolone/eplerenone postdose administration on Day 2/corresponding timepoint for negative control arm.
- Study Arm 3 (Negative Control Arm): no Treatment: Fludrocortisone challenge only Day 1: 1 mg single dose at 9 h predose vamorolone/eplerenone* dosing. Day 2: 0.1 mg and 0.5 mg multiple doses. For detailed timepoints, see protocol Section 4.1. Day 3: 0.1 mg single dose at 24 h postdose vamorolone/eplerenone* dosing.
  *or corresponding timepoint for negative control arm
  Fludrocortisone: Fludrocortisone challenge on Days 1 to 3 (for all subjects):
  Day 1:
  -Fludrocortisone 1 mg at 9 h predose vamorolone /eplerenone administration/corresponding timepoint for negative control arm
  Day 2:
  * Fludrocortisone 0.5 mg at the same time of vamorolone/eplerenone administration in the morning (0 h) /corresponding timepoint for negative control arm.
  * Fludrocortisone 0.1 mg at 2 h, 4 h, 6 h, 8 h, 10 h, 12 h, and 14 h vamorolone/eplerenone postdose administration/corresponding timepoint for negative control arm.
  * Fludrocortisone 0.5 mg at 16 h vamorolone/eplerenone postdose administration/corresponding timepoint for negative control arm.
  Day 3:
  -Fludrocortisone 0.1 mg at 24 h vamorolone/eplerenone postdose administration on Day 2/corresponding timepoint for negative control arm.
Period: Overall Study
Arm/Group | Study Arm 1 (Test Arm)Vamorolone | Study Arm 2 (Positive Control Arm): Eplerenone | Study Arm 3 (Negative Control Arm): no Treatment
Started | 10 | 10 | 10
Completed | 10 | 10 | 10
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Set: All subjects assigned (randomized) to study treatment and received at least 1 dose of study treatment. Subjects were analyzed according to the treatment they received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Arm 1 (Test Arm)Vamorolone | Study Arm 2 (Positive Control Arm): Eplerenone | Study Arm 3 (Negative Control Arm): no Treatment | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.7 (9.91) | 45.3 (10.60) | 35.6 (7.86) | 40.9 (10.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 10 | 10 | 10 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 10 | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 10 | 10 | 10 | 30
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 10 | 10 | 10 | 30
BMI [Mean (Standard Deviation); unit: kg/m2] | 24.69 (3.211) | 26.73 (2.200) | 24.91 (2.295) | 25.44 (2.683)
Weight [Mean (Standard Deviation); unit: kg] | 80.56 (13.828) | 85.45 (13.115) | 78.95 (10.581) | 81.65 (12.465)
Height [Mean (Standard Deviation); unit: cm] | 180.2 (7.44) | 178.3 (6.84) | 177.9 (7.08) | 178.8 (6.95)

OUTCOME MEASURES:

1. Primary Outcome: Determination of the Ratio of Sodium to Potassium (Na/K) in Urine
Description: Amounts of Na and K were calculated by multiplying the respective concentration by the volume of urine for each collection interval. The considered timepoints were:
  Day 1: 24-9 h and 9-0 h predose of vamorolone/eplerenone; Day 2: 0-2 h, 2-4 h, 4-6 h, 6-8 h, 8-10 h, 10-12 h, 12-14 h, 14-16 h, 16-24 h postdose vamorolone/eplerenone or corresponding timepoint for negative control arm with fludrocortisone administrations (no treatment) Day 3: 24-32 h, 32-40 h, 40-48 h postdose vamorolone/eplerenone or corresponding timepoint for negative control arm with fludrocortisone administrations (no treatment)
  The individual Na/K ratio was then calculated for each urine collection interval using the amounts of Na and K. The corresponding logarithm of the Na/K ratio was determined. To avoid negative values, the ratio was multiplied by 10 before transformation, i.e., log10(10*Na/K).
Time Frame: Day 1, Day 2 and Day 3
Population: This set is a subset of the Safety Set and includes all subjects who completed the study without any findings/events likely affecting Pharmacodynamic (PD).
Measure: Geometric Mean (Standard Deviation); unit: log10(10*Na/K)
Arm/Group | Study Arm 1 (Test Arm)Vamorolone | Study Arm 2 (Positive Control Arm): Eplerenone | Study Arm 3 (Negative Control Arm): no Treatment
Number analyzed (Participants) | 10 | 10 | 10
log10(10*Na/K)
  Day 1; 24-9h predose (Baseline) | 1.12929 (1.090602) | 0.98207 (1.290309) | 1.04238 (1.407236)
  Day 1; 9-0h predose | 0.54902 (1.483174) | 0.55352 (1.508765) | 0.45720 (1.788948)
  Day 2; 0-2h postdose | 0.57742 (1.168846) | 0.49927 (1.565160) | 0.53698 (1.351042)
  Day 2; 2-4h postdose | 0.61770 (1.506227) | 0.68844 (1.363715) | 0.47736 (1.297863)
  Day 2; 4-6h postdose | 0.93496 (1.227122) | 0.98531 (1.198851) | 0.20520 (1.715714)
  Day 2; 6-8h postdose | 0.59716 (1.849719) | 1.12174 (1.150301) | 0.31908 (1.543390)
  Day 2; 8-10h postdose | 0.54634 (2.263355) | 1.06596 (1.257710) | 0.23369 (1.627840)
  Day 2; 10-12 h postdose | 0.34996 (2.319486) | 0.57545 (2.918277) | 0.16923 (5.317341)
  Day 2; 12-14h postdose | 0.30144 (3.085968) | 0.61696 (2.726467) | 0.16288 (4.000192)
  Day 2; 14-16h postdose | 0.23802 (1.551328) | 0.63605 (2.092207) | 0.28266 (1.968431)
  Day 2; 16-24h postdose | 0.37176 (1.372678) | 0.34487 (4.249965) | 0.21423 (2.165262)
  Day 3; 24-32h postdose: number analyzed (Participants) | 10 | 09 | 10
  Day 3; 24-32h postdose | 0.81275 (1.231294) | 0.46217 (1.617748) | 0.50869 (1.304142)
  Day 3; 32-40h postdose | 0.79158 (1.432755) | 0.81390 (1.370027) | 0.94041 (1.448171)
  Day 3; 40-48h postdose: number analyzed (Participants) | 10 | 09 | 10
  Day 3; 40-48h postdose | 0.88696 (1.412253) | 1.03802 (1.282118) | 0.98064 (1.250503)

2. Secondary Outcome: Vamorolone PK Parameter AUC0-tlast
Description: The area under the concentration-time curve (AUC) from time zero (= dosing time) to the time of the last quantifiable concentration (tlast). The collection points used to determine the curve were as follows: predose; and 1, 2, 4, 8, 12, 24 h postdose on Day 2
Time Frame: Day 2
Population: This set is a subset of the Safety Set and includes all subjects who completed the study without any findings/events likely affecting PK.
Measure: Mean (Standard Deviation); unit: h*ng/ml
Groups:
- Study Arm 1 (Test Arm): Vamorolone: single oral dose of vamorolone 20 mg/kg on day 2
  + Fludrocortisone Challenge Day 1: 1 mg single dose at 9 h predose vamorolone dosing. Day 2: 0.1 mg and 0.5 mg multiple doses. For detailed timepoints, see protocol Section 4.1. Day 3: 0.1 mg single dose at 24 h postdose vamorolone dosing.
  Vamorolone: vamorolone 20 mg/kg single dose on Day 2
  Fludrocortisone: Fludrocortisone challenge on Days 1 to 3 (for all subjects):
  Day 1:
  -Fludrocortisone 1 mg at 9 h predose vamorolone /eplerenone administration/corresponding timepoint for negative control arm
  Day 2:
  * Fludrocortisone 0.5 mg at the same time of vamorolone/eplerenone administration in the morning (0 h) /corresponding timepoint for negative control arm.
  * Fludrocortisone 0.1 mg at 2 h, 4 h, 6 h, 8 h, 10 h, 12 h, and 14 h vamorolone/eplerenone postdose administration/corresponding timepoint for negative control arm.
  * Fludrocortisone 0.5 mg at 16 h vamorolone/eplerenone postdose administration/corresponding timepoint for negative control arm.
  Day 3:
  -Fludrocortisone 0.1 mg at 24 h vamorolone/eplerenone postdose administration on Day 2/corresponding timepoint for negative control arm.
Arm/Group | Study Arm 1 (Test Arm): Vamorolone
Number analyzed (Participants) | 10
h*ng/ml | 19802.6 (4422.56)

3. Secondary Outcome: Vamorolone PK Parameter AUC0-inf
Description: The AUC from time zero (dosing time) extrapolated to infinity estimated. The collection points used to determine the curve were as follows: predose; and 1, 2, 4, 8, 12, 24 h postdose on Day 2
Time Frame: Day 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*ng/ml
Arm/Group | Study Arm 1 (Test Arm): Vamorolone
Number analyzed (Participants) | 10
h*ng/ml | 19879.8 (4419.77)

4. Secondary Outcome: Vamorolone PK Parameter Cmax
Description: Maximum plasma drug concentration after administration of vamorolone. For this PK measure, the following timepoints were considered: predose; and 1, 2, 4, 8, 12, 24 h postdose on Day 2
Time Frame: Day 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Study Arm 1 (Test Arm): Vamorolone
Number analyzed (Participants) | 10
ng/mL | 3942 (1018.7)

5. Secondary Outcome: Vamorolone PK Parameter Tmax
Description: Time to reach maximum concentration following vamorolone administration. For this PK measure, the following timepoints were considered: predose; and 1, 2, 4, 8, 12, 24 h postdose on Day 2
Time Frame: Day 2
Population: as for outcome 2
Measure: Median (Full Range); unit: h
Arm/Group | Study Arm 1 (Test Arm): Vamorolone
Number analyzed (Participants) | 10
h | 1.992 [1.00 to 2.00]

6. Secondary Outcome: Vamorolone PK Parameter t1/2
Description: Elimination half-life is the amount of time it takes for the concentration of a drug in the body to decrease by half. For this PK measure, the following timepoints were considered: predose; and 1, 2, 4, 8, 12, 24 h postdose on Day 2
Time Frame: Day 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Study Arm 1 (Test Arm): Vamorolone
Number analyzed (Participants) | 10
h | 3.170 (0.6253)

7. Secondary Outcome: Eplerenone PK Parameters AUC0-tlast
Description: The area under the concentration-time curve (AUC) from time zero (= dosing time) to the time of the last quantifiable concentration (tlast).The collection points used to determine the curve were as follows: predose; and 1, 2, 4, 8, 12, 24 h postdose on Day 2
Time Frame: Day 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*ng/ml
Arm/Group | Study Arm 2 (Positive Control Arm): Eplerenone
Number analyzed (Participants) | 10
h*ng/ml | 18631.4 (9242.04)

8. Secondary Outcome: Eplerenone PK Parameter AUC0-inf
Description: The AUC from time zero (dosing time) extrapolated to infinity. The collection points used to determine the curve were as follows: predose; and 1, 2, 4, 8, 12, 24 h postdose on Day 2
Time Frame: Day 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*ng/ml
Arm/Group | Study Arm 2 (Positive Control Arm): Eplerenone
Number analyzed (Participants) | 10
h*ng/ml | 19899.9 (11361.57)

9. Secondary Outcome: Eplerenone PK Parameter Cmax
Description: Maximum plasma drug concentration after administration of eplerenone. For this PK measure, the following timepoints were considered: predose; and 1, 2, 4, 8, 12, 24 h postdose on Day 2
Time Frame: Day 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Study Arm 2 (Positive Control Arm): Eplerenone
Number analyzed (Participants) | 10
ng/ml | 2362 (551.42)

10. Secondary Outcome: Eplerenone PK Parameter Tmax
Description: Time to reach to the maximum concentration after eplerenone. For this PK measure, the following timepoints were considered: predose; and 1, 2, 4, 8, 12, 24 h postdose on Day 2
Time Frame: Day 2
Measure: Median (Full Range); unit: h
Arm/Group | Study Arm 2 (Positive Control Arm): Eplerenone
Number analyzed (Participants) | 10
h | 2.000 [0.97 to 2.02]

11. Secondary Outcome: Eplerenone PK Parameter t1/2
Description: as for outcome 6
Time Frame: Day 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Study Arm 2 (Positive Control Arm): Eplerenone
Number analyzed (Participants) | 10
h | 4.453 (2.2996)

ADVERSE EVENTS:
Time Frame: All adverse events AEs)and serious AE(SAEs) were collected from the signing of the informed consent until the safety follow-up phone call on Day11. All SAEs were to be recorded & reported to the sponsor within 24hours of awareness,filing in the safety form provided. Investigators were not obligated to actively seek AEs or SAEs after conclusion of the study participation. If the investigator learned of any SADR (SAE considered related to the IMP) at any time it had to be reported to the sponsor
Arm/Group | Study Arm 1 (Test Arm)Vamorolone | Study Arm 2 (Positive Control Arm): Eplerenone | Study Arm 3 (Negative Control Arm): no Treatment
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 1/10 | 2/10 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Arm 1 (Test Arm)Vamorolone (N=10) | Study Arm 2 (Positive Control Arm): Eplerenone (N=10) | Study Arm 3 (Negative Control Arm): no Treatment (N=10)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Mild headache was reported approximately 1 hour after vamorolone administration on Day 2 and lasted for 7.5 h. The event resolved without any concomitant medication but was condisered related to vamolorone.
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) — Two mild nasopharyngitis in subjects treated with eplerenone. One with rhinitis and pharyngitis started on Day 7 and resolved in about 4 days. The other started on Day 5 and took about 8 days to resolve. Neither subject took concomitant medication.
Circulatory collaspse (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) — A subject treated with eplerenone experienced moderate circulatory collapse on Day 4, which lasted approximately one hour. This event was not considered to be related to the study treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-02-26): https://cdn.clinicaltrials.gov/large-docs/09/NCT06649409/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-17): https://cdn.clinicaltrials.gov/large-docs/09/NCT06649409/SAP_001.pdf